CLINICAL TRIAL: NCT06419296
Title: Mortality of MBL-producing Enterobacteriaceae Bacteremias with the Combined Use of Ceftazidime-avibactam and Aztreonam Vs. Other Active Antibiotics. a Multicenter Target Trial Emulation.
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Mariana Vaena, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 6915
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Bacteremia
Keywords: multicenter; target trial emulation; bacteremia; metallo-beta-lactamase; carbapenemase-producing Enterobacteriaceae; ceftazidime-avibactam aztreonam
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CAZAVI + ATM: patients who received antibiotic therapy with a standard bacteremia treatment dose of Ceftazidima-Avibactam + Aztreonam (2.5 grams every 8 hours of ceftazidime-avibactam + 2 grams every 8 hours of aztreonam). Dosage adjustments for prolonged infusion or according to renal function will be considered.
- Other Active Antibiotics treatment group: Patients who received a combination or at least one of the following antibiotics, with doses adjusted according to renal function:
  Colistin: 300 mg loading and 150 mg maintenance every 12 hours. Meropenem: 1000 or 2000 mg every 8 hours via infusion in 30 minutes or 3 hours. Fosfomycin: 12 to 24 grams per day, divided every 6 to 8 hours. Aminoglycoside (amikacin: 15 mg/kg/24 hours or gentamicin: 7 mg/kg/24 hours). Tigecycline: 100 or 200 mg loading and 50 or 100 mg maintenance every 12 hours.

SUMMARY:
Ceftazidime-avibactam and aztreonam combination (CAZAVI + ATM) presents a potential alternative for the treatment of metallo-beta-lactamase (MBL)-type carbapenemase-producing Enterobacteriaceae (CPE) bacteremia, particularly where Cefiderocol is not readily available.

This study proposes a Target Trial Emulation (TTE) to assess the efficacy and safety of CAZAVI + ATM compared to other active antibiotics (OAAs) in patients with MBL-type CPE bacteremia, and also to evaluate all-cause 30-day mortality, resistance profiles of isolated microorganisms, clinical failure rates, leukocyte count normalization, adverse events, occurrence of Clostridium difficile infection, and emergence of new multidrug-resistant microorganisms.

Data will be collected through the REDCap database, with rigorous verification for completeness and accuracy.

The outcomes of this project will contribute vital insights into the efficacy and safety of CAZAVI + ATM, informing clinical practice guidelines for the management of MBL-type bacteremia across diverse settings.

DETAILED DESCRIPTION:
Patients will be categorized into two treatment groups for analysis:

CAZAVI + ATM treatment group and Other Active Antibiotics treatment group. As this study is retrospective, treatment group assignment will not be a randomized procedure. Allocation data will be collected from medical records as a dichotomous variable.

In the present study, allocation to CAZAVI + ATM or OAAs will depend on various factors such as drug availability, hospital costs, and medical criteria. Therefore, to ensure comparability among participant characteristics, baseline factors will be adjusted to mitigate indication bias.

To simulate randomization at baseline (identification of MBL-type CPE in blood samples), ensuring comparability between treatment groups, several covariates will be balanced: age, sex, comorbidities (Charlson score), Pitt score, immunosuppression with neutropenia, immunosuppression without neutropenia, days of hospitalization prior to culture, Sequential Organ Failure Assessment (SOFA) score, days of effective antibiotic treatment between blood culture and positivization [25]. Also, as this is a multicenter study, it will be adjusted for the characteristics of the center (public-private), including a total of 10 variables to be adjusted for.

The start of the follow-up period (Time Zero or T0) will be defined by the identification of MBL-type CPE in at least one clinical blood sample (blood culture or PCR). From this point on, all patients will be followed up. A 24-hour grace period will be considered from the identification of MBL-type CPE until the patient initiates either of the two treatment groups.

To mitigate immortality bias, the initiation of both treatment strategies will synchronize with the eligibility criteria at Time Zero of follow-up. Thus, every patient must remain alive from blood culture collection until MBL detection to be eligible for inclusion in the study, and antibiotic treatment must be initiated within 24 hours of detection. All enrolled patients will be followed until 30 days after inclusion in the study, death, or hospital discharge, whichever occurs first.

A sample calculation was performed to test the null hypothesis of equality in the proportion of deaths among patients who received CAZAVI + ATM vs. OAAs. Falcone et al. reported a 19% mortality rate 30 days after inclusion in the CAZAVI + ATM arm and a 44% mortality rate in patients with OAAs. However, for the present study we consider an 80% power is necessary to detect a clinically relevant difference of 15%, therefore we expect a mortality of 34% in the OAAs arm and 19% in the CAZAVI + ATM arm. With an alpha of 5%, two-tailed test, expected ratio CAZAVI + ATM/OAAs of 1:1, a sample size of 270 patients (135 for each branch) is calculated.

Finally, to address indication bias, an adjustment will be made with Propensity Score (PS) matching. Considering 10 confounders entered into the model, at least 10 to 20 events will be required for each variable. Therefore, as the outcome of the PS will be the CAZAVI + ATM exposure variable, at least 150 patients in the CAZAVI + ATM branch will be required. Thus,we consider the calculation of 300 patients, 150 per branch.

A meticulous data collection plan will be carried out to ensure accuracy and confidentiality of the information collected. The following procedures will be implemented:

Data source: Data will be obtained from paper or electronic medical records from each participating center. Patient tracking will be done through the bacteriology records of each hospital center.

Data recording: Variables for each patient will be uploaded to a centralized REDCap database. The principal investigator and associated investigators of each participating center will be responsible for data upload. To maintain privacy and confidentiality, each patient will receive a randomly generated registration number to anonymize their identity in the database.

Data access: Access to center-specific data will be restricted to the principal investigators. Researchers will access REDCap using personal credentials, limiting data access to authorized personnel only.

Confidentiality and anonymization: Adherence to legal provisions, such as the Argentinian National Personal Data Protection (number 25.326) and the Habeas Data, will be strictly complied with in order to protect the confidentiality and privacy of the patients involved in the study. All collected data will be anonymized, devoid of patient identifiers.

Data storage: Once the data upload is completed, the entire database will be stored under password and will only be available to the principal investigators of the study. All necessary precautions will be taken to ensure that the data are maintained in a secure and reliable environment.

The research team is dedicated to upholding data privacy, complying with legal regulations, and conducting the study ethically and responsibly.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Confirmed bacteremia by MBL-type Carbapenemase-Producing Enterobacteriaceae (CPE)
* Initiation of effective antibiotic therapy within 24 hours of identification of MBL-type CPE and within 96 hours of blood sample.

Exclusion Criteria:

* Bacteremia due to the following complicated infections:

  * Endocarditis or other endovascular infection without extractable focus.
  * Necrotizing fasciitis
  * Osteomyelitis or septic arthritis
  * Confirmed prostatitis
  * Non-drainable abscess or other unresolved infection requiring surgical intervention (e.g., cholecystitis)
  * Central nervous system infections
  * Empyema
* Successive episodes of bacteremia by the same pathogen (with the same resistance profile) within the previous 60 days.
* Polymicrobial bacteremias, not classified as contaminants.
* Patients with documented allergy to beta-lactams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include a cohort of hospitalized patients from Argentine hospitals. Hospital centers will be invited to participate through the network of the Argentine Society of Medicine (SAM), the Argentine Society of Intensive Care (SATI) and the Argentine Society Of Infectious Diseases (SADI).
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | within 30 days from the initiation of treatment (follow-up period)
  death from any cause

SECONDARY OUTCOMES:
Describe the resistance profile of the isolated microorganisms | 30-day follow-up period
  including the associated enzymatic mechanisms
Compare clinical failure | 30-day follow-up period
  presence of 1) Relapse: recurrent bacteremia due to the same bacteria; 2) Restart of antibiotic therapy targeting the same germs; 3) Local suppurative complication that was not present at the beginning of the infection; 4) Distant complications of the initial infection (defined by the growth of the same bacteria causing the initial bacteremia in distant sites)
Compare the number of days to normalization of the leukocyte count in the laboratory | 30-day follow-up period
  (leukocyte count less than 12x109/L). (leukocyte co(leukocyte count less than 12x109/L).unt less than 12x109/L)
Compare the proportion of adverse events | 30-day follow-up period
  including: neutropenia, thrombocytopenia, renal failure, hepatotoxicity, skin reactions and ion-losing tubulopathy
compare the occurrence of Clostridium difficile infection | 30-day follow-up period
  Appearance of positive C. difficile toxin or positive C. difficile PCR
compare the occurrence of new multidrug-resistant microorganisms | 30-day follow-up period
  such as KPC, NDM, VIM, IMP, OXA or EVR-producing CLD, detected in both clinical and surveillance samples

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Huespe, MD, MPh, Study Director — Hospital Italiano de Buenos Aires
Locations (16):
- Argentina (16):
  - Hospital Municipal de Agudos Dr. Leónidas Lucero, Bahía Blanca, Buenos Aires
  - Hospital Interzonal General de Agudos ''Profesor Dr. Luis Güemes'', Haedo, Buenos Aires
  - Hospital de Alta Complejidad del Bicentenario Esteban Echeverria, Monte Grande, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Municipal Central de San Isidro "Dr. Melchor Ángel Posse", San Isidro, Buenos Aires
  - Hospital Presidente Perón, Sarandí, Buenos Aires
  - Sanatorio Franchin, Buenos Aires, Buenos Aires F.D.
  - Hospital Alemán, Buenos Aires, Buenos Aires F.D.
  - Hospital de Infecciosas Francisco Javier Muñiz, Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Hospital Médico Policial Churruca Visca, Buenos Aires, Buenos Aires F.D.
  - Hospital Privado Universitario de Córdoba, Córdoba, Córdoba Province
  - Hospital Interdistrital Evita, Formosa, Formosa Province
  - Hospital Italiano Rosario, Rosario, Santa Fe Province
  - Hospital José Bernardo Iturraspe, Santa Fe, Santa Fe Province
  - Hospital José María Cullen, Santa Fe, Santa Fe Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] al-Hasany M, Mohamed AS. Veno-occlusive disease of the liver in Iraq. Nine cases occurring in three Bedouin families. Arch Dis Child. 1970 Oct;45(243):722-4. doi: 10.1136/adc.45.243.722. No abstract available. PMID 5477705
- [Background] Zhou R, Fang X, Zhang J, Zheng X, Shangguan S, Chen S, Shen Y, Liu Z, Li J, Zhang R, Shen J, Walsh TR, Wang Y. Impact of carbapenem resistance on mortality in patients infected with Enterobacteriaceae: a systematic review and meta-analysis. BMJ Open. 2021 Dec 14;11(12):e054971. doi: 10.1136/bmjopen-2021-054971. PMID 34907071
- [Background] Lee YL, Ko WC, Hsueh PR. Geographic patterns of global isolates of carbapenem-resistant Klebsiella pneumoniae and the activity of ceftazidime/avibactam, meropenem/vaborbactam, and comparators against these isolates: Results from the Antimicrobial Testing Leadership and Surveillance (ATLAS) program, 2020. Int J Antimicrob Agents. 2022 Nov-Dec;60(5-6):106679. doi: 10.1016/j.ijantimicag.2022.106679. Epub 2022 Oct 12. PMID 36241011
- [Background] Morey LC, Blashfield RK. Empirical classifications of alcoholism: a review. J Stud Alcohol. 1981 Nov;42(11):925-37. doi: 10.15288/jsa.1981.42.925. No abstract available. PMID 7038311
- [Background] El Nekidy WS, Al Ali M, Abidi E, Ghazi IM, Attallah N, El Lababidi R, Mooty M, Ghosn M, Mallat J. Microbiologic outcomes of ceftazidime-avibactam dosing in patients with sepsis utilizing renal replacement therapies. Hemodial Int. 2023 Jul;27(3):289-295. doi: 10.1111/hdi.13090. Epub 2023 May 5. PMID 37144742
- [Background] Caston JJ, Cano A, Perez-Camacho I, Aguado JM, Carratala J, Ramasco F, Soriano A, Pintado V, Castelo-Corral L, Sousa A, Farinas MC, Munoz P, Abril Lopez De Medrano V, Sanz-Pelaez O, Los-Arcos I, Gracia-Ahufinger I, Perez-Nadales E, Vidal E, Doblas A, Natera C, Martinez-Martinez L, Torre-Cisneros J. Impact of ceftazidime/avibactam versus best available therapy on mortality from infections caused by carbapenemase-producing Enterobacterales (CAVICOR study). J Antimicrob Chemother. 2022 Apr 27;77(5):1452-1460. doi: 10.1093/jac/dkac049. PMID 35187577
- [Background] Lafrance C, Dumont M, Lesperance P, Lambert C. Daytime vigilance after morning bright light exposure in volunteers subjected to sleep restriction. Physiol Behav. 1998 Mar;63(5):803-10. doi: 10.1016/s0031-9384(97)00538-6. PMID 9618002
- [Background] Qu J, Xu J, Liu Y, Hu C, Zhong C, Lv X. Real-world effectiveness of ceftazidime/avibactam versus polymyxin B in treating patients with carbapenem-resistant Gram-negative bacterial infections. Int J Antimicrob Agents. 2023 Aug;62(2):106872. doi: 10.1016/j.ijantimicag.2023.106872. Epub 2023 May 27. PMID 37247645
- [Background] Jacobson BH, Aldana SG, Goetzel RZ, Vardell KD, Adams TB, Pietras RJ. The relationship between perceived stress and self-reported illness-related absenteeism. Am J Health Promot. 1996 Sep-Oct;11(1):54-61. doi: 10.4278/0890-1171-11.1.54. PMID 10163451
- [Background] Matsui I, Yoneda S, Ishikawa K, Miyairi S, Fukui S, Umeyama H, Honda K. Roles of the aromatic residues conserved in the active center of Saccharomycopsis alpha-amylase for transglycosylation and hydrolysis activity. Biochemistry. 1994 Jan 18;33(2):451-8. doi: 10.1021/bi00168a009. PMID 8286375
- [Background] Royer P. [Genetics and nephropathies]. Rev Fr Etud Clin Biol. 1969 Nov;14(9):839-42. No abstract available. French. PMID 5365724
- [Background] Falcone M, Daikos GL, Tiseo G, Bassoulis D, Giordano C, Galfo V, Leonildi A, Tagliaferri E, Barnini S, Sani S, Farcomeni A, Ghiadoni L, Menichetti F. Efficacy of Ceftazidime-avibactam Plus Aztreonam in Patients With Bloodstream Infections Caused by Metallo-beta-lactamase-Producing Enterobacterales. Clin Infect Dis. 2021 Jun 1;72(11):1871-1878. doi: 10.1093/cid/ciaa586. PMID 32427286
- [Background] Marks LE, Wheeler ME. Attention and the detectability of weak taste stimuli. Chem Senses. 1998 Feb;23(1):19-29. doi: 10.1093/chemse/23.1.19. PMID 9530966
- [Background] Huttner A, Albrich WC, Bochud PY, Gayet-Ageron A, Rossel A, Dach EV, Harbarth S, Kaiser L. PIRATE project: point-of-care, informatics-based randomised controlled trial for decreasing overuse of antibiotic therapy in Gram-negative bacteraemia. BMJ Open. 2017 Jul 13;7(7):e017996. doi: 10.1136/bmjopen-2017-017996. PMID 28710229
- [Background] Tingsgard S, Bastrup Israelsen S, Ostergaard C, Benfield T. Emulating a Target Trial of Shorter Compared to Longer Course of Antibiotic Therapy for Gram-Negative Bacteremia. Clin Infect Dis. 2024 Feb 17;78(2):292-300. doi: 10.1093/cid/ciad670. PMID 37949816
- See also: Global antimicrobial resistance and use surveillance system (GLASS) report: 2022. World Health Organization; 9 Dec 2022 [cited 3 Oct 2023]. — https://www.who.int/publications/i/item/9789240062702
- See also: Surveillance of antimicrobial resistance in Europe 2017. In: European Centre for Disease Prevention and Control — https://www.ecdc.europa.eu/en/publications-data/surveillance-antimicrobial-resistance-europe-2017